CLINICAL TRIAL: NCT03477513
Title: Personalized Treatment of Glioblastoma Via Image-Guided Predictive Modeling of Recurrence: A Single-Arm, Single Institutional Pilot Prospective Study of Dose-Escalated Radiation Therapy
Brief Title: Personalized Radiation Therapy for GBM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 24317
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Dose-escalated radiation therapy
  Interventions: Radiation: Radation Therapy

INTERVENTIONS:
Radiation: Radation Therapy — Personalized Radiation Therapy

SUMMARY:
The study is a pilot study to estimate the efficacy of personalized dose-escalation radiation therapy in patients with glioblastoma, as measured by estimating the median of progression-free survival. Toxicity, patterns of recurrence, and overall median survival will be measured as secondary endpoints. Adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven WHO Grade IV glioblastoma, after gross-total or near-total resection, who are undergoing definitive chemoradiation as part of their treatment regimen
* Age 18 or older
* Ability to give signed informed consent
* Karnofsky Performance Status (KPS) at least 70

Exclusion Criteria:

* Placement of Gliadel wafers
* Participation in another investigational trial
* Active treatment of another malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Alonso-Basanta, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided